CLINICAL TRIAL: NCT06187155
Title: Impact of Education Level on Clinical Outcomes in Self-INR Managed Patients on Longterm Warfarin: a Single-center Randomized Controlled Study
Brief Title: Impact of Education Level on Clinical Outcomes in Self-INR Managed Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Collaborators: Magdi Yacoub Heart Foundation (Other)
Responsible Party: Principal Investigator, Hossameldin Elsayed Khalifa Hussein, Associate Specialist of Adult Cardiology, Magdi Yacoub Heart Foundation
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 20230614MYFAHC_INR
Record Dates: First submitted 2023-12-16; First posted 2024-01-02 (Actual); Last update posted 2024-09-05 (Actual); Status verified 2024-08

CONDITIONS: Atrial Fibrillation and Flutter; Mechanical Mitral Valve Prosthesis
Keywords: INR self-management; education level; warfarin; time in therapeutic range
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- INR-self management (Experimental): The participants will be responsible to monitor their INR regularly and adjust the warfarin dose by themselves accordingly, without seeking medical advice from medical personnel for 6 months.
  All participants will receive full education class of minimum one-hour time and training about how to interpret INR levels and adjust their medication dose according to a pre-determined dose-INR schedule.
  Interventions: Other: INR self-management
- Standard of care (No Intervention): Regular INR monitoring and seeking medical advice at Aswan Heart Centre

INTERVENTIONS:
Other: INR self-management — will receive full education class of minimum one-hour time and training about how to interpret INR levels independently and adjust their medication dose according to a pre-determined dose-INR schedule.
  Arms: INR-self management

SUMMARY:
Oral anticoagulation (OAC) is indicated in a wide variety of clinical conditions including atrial fibrillation (AF), mechanical valve prosthesis (MVP), deep vein thrombosis and pulmonary embolism. Although direct OAC has replaced vitamin K antagonists (VKA) in non-valvular AF due to lower bleeding risk, it's still recommended to use VKA specifically in cases of valvular AF, MVP and anti-phospholipid syndrome.

VKA has a narrow therapeutic range and multiple drug interactions causing unpredicted pharmacodynamics. This requires regular monitoring of the international normalized ratio (INR) level to ensure it's in the target therapeutic range and prevent extreme values that may result in thrombo-embolic events or sometimes fatal bleeding.

Self-INR monitoring and management have emerged recently as a safe cost-effective alternative to standard management, with evidence of tighter control of INR, reduction of thrombo-embolic events, and improving treatment-related quality of life. However, there are no specific criteria for patient selection. Whether the level of education and other social factors would affect the outcomes of self-management is still not clear.

Owing to the wide geographical area served by Aswan Heart Center, many patients have to cover long distances to follow up their INR and seek medical advice regarding adequate dose modification. This may result in reluctance and non-compliance to clinic visits and INR testing. Proper education, training and providing an alternative near place to measure the INR and self-adjust warfarin dose is expected to improve patient adherence and compliance.

DETAILED DESCRIPTION:
Study Methods

* Population of study: Patients who have a clinical indication for long term VKA.
* Study location: Aswan Heart Center.
* Inclusion criteria: Adult patients above 18 years who are indicated for long term VKA and has been on VKA for more than 6 months.
* Exclusion criteria:

  1. Refusal to join the study. 2. History of life-threatening bleeding or thrombo-embolic events. 3. Illiterate patients with no caregivers living at the same home.
* Patient informed consent:

Individual informed consent will be taken from every candidate for the study. The candidates will have the right to withdraw from the study at any time without any changes in the clinical service provided to them.

- Methodology in details:

A-Medical history including:

Age, gender, indication of VKA. Data about valve surgery including date, location and type of valve. Past history of any chronic medical conditions, thrombo-embolic or bleeding events. Past history of blood transfusion.

B-Social history including:

Marital status, occupation, level of education and self-care capability.

C- Clinical examination including:

Assessment of body weight, height and body mass index calculation. Vital signs including blood pressure measurement using standard technique, assessment of the pulse, respiratory rate and temperature.

C- Blood sample and chemistry:

Blood tests will be done for all participants initially and at the end of the study. Laboratory workup will include complete blood count, liver, kidney function tests and electrolytes.

F- Electrocardiography (ECG):

12-lead ECG will be done for all participants initially and the end of the study to confirm rhythm.

H- Echocardiography:

* Trans-thoracic echocardiography will be done for all patients to assess valve function, leaflet excursion, peak and mean pressure gradients across the valve.
* In case of abnormally elevated pressure gradients, abnormal leaflet motion or suspected prosthesis-related mass, trans-oesophageal echocardiography will be done to confirm or exclude MVP malfunction.

I. Randomization:

* Patients will be randomized with the ratio of 1:1 to undergo self-management of INR versus standard management in the anticoagulation clinic using a randomization table.
* Self-management arm:

  • All participants will receive full education class of minimum one-hour time and training about how to interpret INR levels and adjust their medication dose according to a pre-determined dose-INR schedule.

  • A registered nurse will be responsible for education and training. Another registered nurse would be responsible to check the participant feedback and well-understanding.

  • The participant will receive a chart to record INR results, test dates and dose modifications for the upcoming 6 months.

  • The participant will be educated about bleeding events, how to grade and when to seek medical attention immediately.

  • The participant will be educated about early manifestations of thrombo-embolism including shortness of breath, focal neurological deficits or lower limb pain.

  • If INR exceeds 8 at any time, the participant will be instructed to urgently contact the center and seek medical advice, he/she will be withdrawn from the trial and switched to the standard monitoring care.

  • If major bleeding or thrombotic event occurred, the participant will be instructed to contact us urgently and will be withdrawn from the trial and switched to the standard monitoring care.
* Standard monitoring arm:

  * This group will be managed according to the local protocol of INR monitoring in a dedicated anticoagulation clinic. A registered nurse (supervised by a physician) would be responsible for medication dose adjustment, scheduling tests and recording any thrombo-embolic or bleeding events.

K. Follow-up:

Standard monitoring group will be reviewed on monthly basis or less according to INR test results. Self-management group will be reviewed 6 months after randomization, with the following data to be obtained:

1. All-cause death.
2. Bleeding events will be graded according to BARC classification

   * Minor bleeding Type 1: self-controlled bleeding that doesn't need seeking medical advice.
   * Major bleeding Type 2: Overt bleeding that requires medical intervention or hospitalization. Type 3a: Bleeding with Hb drop (3-5 gm/dL), or requiring blood transfusion. Type 3b: Bleeding with Hb drop 5 gm/dL or more, or requiring surgical intervention.

Type 4: Coronary artery bypass graft-related bleeding. Type 5: Fatal bleeding. 4. Thrombo-embolic event: defined as mechanical valve thrombosis confirmed by trans-oesophageal echocardiography (prosthesis-related mass, elevated gradients, stuck leaflet motion), cerebrovascular stroke, peripheral embolism causing acute limb ischemia.

5. Time and proportion of tests in therapeutic range will be calculated using Rosendaal method.

6. Frequency of tests will be recorded.

In case of mortality, data will be collected about the date and cause of mortality, and any reported clinical events before mortality.

Data will be presented and used without inference to the name or personal data of the patients. All patient records will be handled in accordance to hospital and national confidentiality protocols.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients above 18 years who are indicated for long term VKA and has been on VKA for more than 6 months.

Exclusion Criteria:

1. Refusal to join the study.
2. History of prior life-threatening bleeding or thrombo-embolic events.
3. Illiterate patients with no caregivers living at the same home.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 586 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Time and proportion of INR in therapeutic range | 6 months
  Time in therapeutic range and percentage of test results in therapeutic range

SECONDARY OUTCOMES:
All-cause mortality | 6 months
  Death from any cause
Thrombo-embolic events | 6 months
  Stroke, valve thrombosis or peripheral embolism
Major bleeding | 6 months
  Overt bleeding that requires medical intervention or hospitalization
Minor bleeding | 6 months
  Self-controlled bleeding that doesn't need seeking medical advice
Frequency of testing | 6 months
  Number of tests per specific time range

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Hosny, MD, Study Director — Aswan Heart Centre
Locations (1):
- Aswan Heart Centre, Aswān, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF, CSR